CLINICAL TRIAL: NCT04564014
Title: A Randomized Controlled Trial of an Internet-based Self-help Skill Strengthening (ISSS) Selective Intervention for Secondary School Teachers With Emotional Problems
Brief Title: Internet-based Self-help Skill Strengthening (ISSS) for Secondary School Teachers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Xue YANG, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17180791
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISSS Intervention (Experimental): The intervention group will receive 5 weekly ISSS sessions in addition to the information about mental health, depression, anxiety and available treatment and community resources also recived by the control group.
  Interventions: Behavioral: ISSS; Other: Education Materials
- Wait-list control group (Active Comparator): Members will receive information about mental health, depression, anxiety and available treatment and community resources but not ISSS during the intervention period.
  Interventions: Behavioral: ISSS; Other: Education Materials

INTERVENTIONS:
Behavioral: ISSS — The ISSS aims to help participants acquire problem-solving (e.g., interpersonal problems) and time management based on the treatment manual of the therapy. Video introductions for each session and example teacher characters who depict the targeted problems and demonstrate implementation of coping/management techniques in a variety of situations. ISSS will use metaphors, daily examples, and lively narrative stories to enhance motivation for participation and understanding of the intervention contents. Session 2-5 will assign exercise and homework. Within 48 hours, participants will receive personalized written feedback (e.g., suggestions) from an e-Coach on the exercises they have completed. Participants can contact e-Coaches via the online system if they have any questions regarding the contents. Questions that beyond the contents will be referred to the health psychologist (PI) by e-Coaches.
Other: Education Materials — Participants will recieve education materials addressing the following issues: (1) introduction to mental health and mental illness; (2) signs and symptoms of depression; (3) treatment of depression and available community resources; (4) signs and symptoms of anxiety; (3) treatment of anxiety and available community resources. The education materials will be carefully developed by the health psychologists and clinical psychologist of the research team who are very experienced in education intervention for mental and emotional health.

SUMMARY:
This RCT develops an ISSS program for secondary teachers. The primary objective is to assess the efficacy of such an intervention in reducing depression/anxiety, compared with a WLC group.

DETAILED DESCRIPTION:
Secondary teachers are under great stress and have prevalent mental/emotional health problems with limited coping resources and treatment. Selective intervention with an ISSS program is potentially useful as it is effective in preventing clinical/severe mental disorders and enhancing cost-effectiveness in health promotion.

Objective: This randomized controlled trial (RCT) develops an Internet-based guided self-help intervention for secondary school teachers. The primary objective is to evaluate the relative efficacy of an Internet-based self-help skill strengthening (ISSS) program in reducing levels of depression and/or anxiety among secondary school teachers that have depressive symptoms and anxiety symptoms versus a wait-list control (WLC) group at post-treatment time and the 6-month follow-up.

Subjects and methods: The study design is two-armed RCT. The participants are secondary school teachers (n=427) with at least mild levels of depression ( Patient Health Questionnaire score >=15) and/or anxiety(Generalized Anxiety Disorder score>=20) identified through screening. Evaluation involves surveys at baseline, end of intervention, and 6 months afterwards. In addition to information received by the wait-list control group, the intervention group receives a carefully designed ISSS program with 5 sessions. The control group will participate in the ISSS program after the 6-month follow-up. Trained e-Coaches with a master degree in psychology or counseling will support and provide feedback to the participants.

Outcomes and measures: The primary outcomes are depression and anxiety. Secondary outcomes include perceived stress, self-efficacy, job performance and well-being. Measures of potential mediators (problem-solving and time management) include: the General Self-Efficacy Scale (GSE),the Performance Maintenance Scale (PMS), the World Health Organization Well-Being Index (WHO-5), theProblem Solving Inventory (PSI), and the Time Management Behavior Scale (TMBS).

Data analysis: Intention-to-treat (ITT) analysis will be performed. ANOVA and Chi-square tests will be conducted to test between-group differences in baseline characteristics. Pearson's correlation analyses will be used to test inter-correlations among all outcome variables and mediators. ANCOVA will be used to test changes in outcome variables at post-test or follow-up with pre-scores controlled. Mean improvement scores will be computed by calculating Cohen's d for ISSS as compared to WLC. Remission rates will be calculated (based on percentage of individuals dropping below PHQ-9 and/or GAD-7 cut-offs). Binary logistic regression will be used for odds ratios between the remission rates in ISSS with WLC. PHQ and GAD will be compared in two groups using ANCOVA. Post-test/follow-up score will be compared among two conditions, with pre-scores as covariates, to examine the group effect. The potential mediation effects of problem solving and time management between intervention conditions and emotional problems will be tested by using Structural Equation Modeling (SEM) and bootstrapping analysis.

Implications: The findings may lead to an evidence-based selective intervention online program for the improvement of secondary teachers' mental/emotional health, a problem with scare coping resources and treatment. Enhancement of teachers' mental/emotional health, related knowledge and coping ability (problem solving, time management) would also benefit students.

ELIGIBILITY:
Inclusion Criteria:

* being local Secondary school teachers
* being able to read and understand Chinese
* having access to the Internet
* 9-item Patient Health Questionnaire (PHQ) and/or 7-item Generalized Anxiety Disorder (GAD) score >=5

Exclusion Criteria:

* currently taking psychotropic medication
* being actively suicidal (as measured by item 9 of the PHQ with score >2)
* having severe depression/anxiety (PHQ>=15/GAD score>=20)
* being international Secondary school teachers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-06-09 (Estimated); Study Completion 2023-06-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline depression immediately after the interventions | immediately after the interventions
  The outcome will be measured by the Patient Health Questionnaire (PHQ) consisting of nine questions designed to correspond to the nine diagnostic criteria for major depressive disorder covered in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Items are rated from 0 to 3 according to increased frequency of experiencing difficulties in each area covered. Scores are summed and can range from 0 to 27. Score 10 is often recommended as the cut-off score to detect major depressive disorder. Scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively. The Chinese version has been validated.
Change from baseline depression six months after the interventions] | six months after the interventions]
  The outcome will be measured by the Patient Health Questionnaire (PHQ) consisting of nine questions designed to correspond to the nine diagnostic criteria for major depressive disorder covered in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Items are rated from 0 to 3 according to increased frequency of experiencing difficulties in each area covered. Scores are summed and can range from 0 to 27. Score 10 is often recommended as the cut-off score to detect major depressive disorder. Scores of 5, 10, 15, and 20 represent cut-off points for mild, moderate, moderately severe, and severe depression, respectively. The Chinese version has been validated.
Change from baseline anxiety immediately after the interventions | immediately after the interventions
  The outcome will be measured by the generalized Anxiety Disorder Scale (GAD) is a 7-item instrument developed to identify likely cases of generalized anxiety disorder in primary care patients and it is a widely-used screening tool of anxiety. Items are rated for the last two weeks, using a four-point rating scale for duration from 1 ("not at all") to 5 ("nearly every day").
  A score of 10 or greater represents a cut point for identifying cases of generalized anxiety disorder, while cut points of 5, 10, 15, and 20 are interpreted as representing mild, moderate, moderately severe, and severe levels of anxiety. The Chinese version has been validated.
Change from baseline anxiety at 6 months | six months after the interventions]
  The outcome will be measured by the generalized Anxiety Disorder Scale (GAD) is a 7-item instrument developed to identify likely cases of generalized anxiety disorder in primary care patients and it is a widely-used screening tool of anxiety. Items are rated for the last two weeks, using a four-point rating scale for duration from 1 ("not at all") to 5 ("nearly every day").
  A score of 10 or greater represents a cut point for identifying cases of generalized anxiety disorder, while cut points of 5, 10, 15, and 20 are interpreted as representing mild, moderate, moderately severe, and severe levels of anxiety. The Chinese version has been validated.

CONTACTS AND LOCATIONS:
Overall Officials: Xue Yang, PhD, Principal Investigator — JC School of Public Health and Primary Care, Faculty of Medicine, CUHK
Locations (1):
- Man Kwan QualiEd College, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No